CLINICAL TRIAL: NCT04240613
Title: Tension-free Vaginal Tape Obturator for the Treatment of Urinary Incontinence - Efficacy and Patient Satisfaction in Long-term Follow-up
Brief Title: Tension-free Vaginal Tape Obturator for the Treatment of Urinary Incontinence -Long-term Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13533
Record Dates: First submitted 2020-01-02; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Urinary Incontinence,Stress; Urinary Incontinence, Urge
Keywords: TVT-O; long-term follow-up; retrospective
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- women treated by TVT-O (Other): All women treated by TVT-O during the years this study was made were included.
  Interventions: Device: TVT-O

INTERVENTIONS:
Device: TVT-O — TVT-O is one of the most popular treatments for urinary incontinence (UI). Its efficacy is well established in patients with pure stress urinary incontinence (SUI). Data reporting long-term outcomes of TVT-O for the treatment of mixed urinary incontinence (MUI) or recurrent SUI is scarce. The objective of this study was to evaluate the efficacy and safety and overall patient satisfaction of TVT-O in different subgroups of UI in a long-term follow-up.

SUMMARY:
The efficacy of TVT-O (tension-free vaginal tape obturator) is well established in patients with stress urinary incontinence (SUI). The objective of this study was to evaluate the efficacy, safety and patient satisfaction of TVT-O in patients suffering from primary, mixed (MUI) or recurrent urinary incontinence (UI) in long-term follow-up.

DETAILED DESCRIPTION:
The long-term results after TVT-O have been scarce. At five years no significant differences were seen between TVT (tension-free vaginal tape) and TVT-O for female SUI in a randomized trial. In two studies the patients were followed-up for ten years after the TVT-O procedure. The first randomized study reporting long term outcomes of TVT-O and outside-in TOT (transobturator tape) in women with urodynamic mixed urinary incontinence (MUI) showed that transobturator tension-free vaginal tapes are associated with a good and sustained patient-reported success rate.

The success of the incontinence procedures should be assessed not only with objective measures but also with methods evaluating subjective satisfaction. The aim of this study was to evaluate the efficacy, safety and overall patient satisfaction of the TVT-O technique in a long-term follow-up of patients suffering from primary or recurrent SUI or MUI.

ELIGIBILITY:
Inclusion Criteria:

We included all the patients who underwent the TVT-O operation between August 2004 and October 2011 in our hospital, Turku university hospital Finland.

Exclusion Criteria:

No exclusion criteria were applied.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — TVT-O is only for females, to treat female urinary incontinence.
Enrollment: 106 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
objective and subjective treatment success | 9.25 years
  Objective treatment success was a negative cough stress test (CST), The CST was performed with a bladder volume of 300 ml aiming on adjusting the tape to allow a drop of saline to escape from the outer meatus of the urethra on strong coughing. The patient was subjectively cured if she answered to being very satisfied or satisfied with the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Eija Laurikainen, Study Director — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No